CLINICAL TRIAL: NCT03621189
Title: The Impacts of Theta-burst Stimulation Over Posterior Superior Temporal Sulcus on Children and Adolescents With Autism Spectrum Disorder
Brief Title: The Impacts of Theta-burst Stimulation on Children and Adolescents With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201509413A0
Record Dates: First submitted 2018-07-07; First posted 2018-08-08 (Actual); Results first posted 2021-08-27 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2018-08

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active-Active (Active Comparator): Participants received the real intervention of TBS (iTBS 1200) over the posterior superior temporal sulcus for 8 weeks (2 days/week).
  *iTBS = intermittent theta burst stimulation
  Interventions: Device: intermittent theta burst stimulation
- Sham-Active (Sham Comparator): Participants received the sham intervention of TBS (coil tilted one-wing 90° off the head) over the posterior superior temporal sulcus for 4 weeks (2 days/week) and then received the real intervention of TBS (iTBS 1200) over the posterior superior temporal sulcus for 4 weeks (2 days/week).
  *iTBS = intermittent theta burst stimulation
  Interventions: Device: intermittent theta burst stimulation

INTERVENTIONS:
Device: intermittent theta burst stimulation — stimulatory protocol

SUMMARY:
The investigator would like to investigate the impact of theta-burst stimulation over posterior superior temporal sulcus in children and adolescents with autism spectrum disorder

ELIGIBILITY:
Inclusion Criteria:

* autism spectrum disorder, confirmed by ADOS

Exclusion Criteria:

* current and past systemic disease
* current and past major psychiatric disorders including schizophrenia, bipolar affective disorder and major depressive disorder
* current and past brain injuries
* intelligence < 70
* seizure history
* pregnant

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2016-11-02 (Actual); Primary Completion 2019-04-17 (Actual); Study Completion 2019-04-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ni HC, Chao YP, Tseng RY, Wu CT, Cocchi L, Chou TL, Chen RS, Gau SS, Yeh CH, Lin HY. Lack of effects of four-week theta burst stimulation on white matter macro/microstructure in children and adolescents with autism. Neuroimage Clin. 2023;37:103324. doi: 10.1016/j.nicl.2023.103324. Epub 2023 Jan 7. PMID 36638598

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the total 80 patients, 5 withdrew from the study.
Period: Overall Study
Arm/Group | Active-Active | Sham-Active
Started | 40 | 40
Completed | 40 | 35
Not Completed | 0 | 5
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Physician Decision | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active-Active | Sham-Active | Total
Number analyzed (Participants) | 40 | 35 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 13 (2.8) | 12.5 (2.9) | 12.8 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 35 | 30 | 65
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Full scale intelligence [Mean (Standard Deviation); unit: units on a scale] — Wechsler Adult Intelligence Scale IV can measure the general intelligence with the range from 40-160. The higher scores stand for better intelligence.
  units on a scale | 88.2 (16.7) | 90 (14.7) | 89 (15.8)
Social Responsiveness Scale [Mean (Standard Deviation); unit: units on a scale] — Social Responsiveness Scale can measure the autism clinical severity with the range from 65-260. The lower scores stand for better social responsiveness.
  units on a scale | 107.3 (24) | 102.1 (23.2) | 104.9 (23.8)
Repetitive Behavior Scale-Revised [Mean (Standard Deviation); unit: units on a scale] — RBS-R is a questionnaire that focuses on repetitive behavior. The score ranges from 0-129. The lower scores stand for lower repetitive behavior.
  units on a scale | 32.2 (18.9) | 33.5 (20.6) | 32.8 (19.7)
Eye task [Mean (Standard Deviation); unit: units on a scale] — An advanced test for Theory of Mind. 43 questions in total, the more correct questions stand for better social skills (The score ranges from 0-43).
  units on a scale | 20.8 (8) | 24.8 (6.9) | 22.7 (7.8)
Frith-Happe Animation (Total) [Mean (Standard Deviation); unit: units on a scale] — A quick and objective test of Theory of Mind. 8 questions in total, the more correct questions stand for better Social Cognition (The score ranges from 0-8).
  units on a scale | 5.5 (2.1) | 5.6 (1.9) | 5.5 (2)
Comorbidity with ADHD [Count of Participants; unit: Participants] | 22 | 14 | 36
Medication (Methylphenidate) [Count of Participants; unit: Participants] | 14 | 10 | 24
Medication (Atomoxetine) [Count of Participants; unit: Participants] | 1 | 1 | 2
Medication (Antipsychotics) [Count of Participants; unit: Participants] | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Changes of Total Scores of Social Responsiveness Scale
Description: Social Responsiveness Scale can measure the autism clinical severity with the range from 65-260. The lower scores stand for better social responsiveness.
Time Frame: baseline; during TBS (4 weeks after baseline); post TBS (8 weeks after baseline); One month follow up (4 weeks after post TBS)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active-Active | Sham-Active
Number analyzed (Participants) | 40 | 35
score on a scale
  Baseline | 107.3 (24) | 102.1 (23.2)
  During TBS | 103.4 (25.5) | 100.1 (27.1)
  Post TBS | 98.5 (28.7) | 95.1 (25.7)
  One month follow up | 97.2 (25.6) | 94.7 (27.9)

2. Primary Outcome: Changes of Total Scores of Repetitive Behavior Scale-Revised
Description: RBS-R is a questionnaire that focuses on repetitive behavior. The score range from 0-129. The lower scores stand for lower repetitive behavior.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active-Active | Sham-Active
Number analyzed (Participants) | 40 | 35
score on a scale
  Baseline | 32.2 (18.9) | 33.5 (20.6)
  During TBS | 28.9 (20.1) | 28.1 (21.5)
  Post TBS | 25.9 (20.5) | 31.5 (23.9)
  One month follow up | 24.3 (17.6) | 29 (23.9)

3. Secondary Outcome: Changes in Accuracy of Frith-Happe Animation
Description: A quick and objective test of Theory of Mind. 8 questions in total, the more correct questions stand for better Social Cognition (The score ranges from 0-48).
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active-Active | Sham-Active
Number analyzed (Participants) | 40 | 35
score on a scale
  Baseline | 5.5 (2.1) | 5.6 (1.9)
  During TBS | 5.4 (1.8) | 5.7 (2.2)
  Post TBS | 5.4 (2) | 5.4 (2.3)
  One month follow up | 5.4 (2.1) | 5.2 (2.6)

4. Secondary Outcome: Changes in Accuracy of Eyes Task
Description: An advanced test for Theory of Mind. 43 questions in total, the more correct questions stand for better social skills (The score ranges from 0-43).
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Sham Control: Participants received the sham intervention of TBS (coil tilted one-wing 90° off the head) over the posterior superior temporal sulcus for 4 weeks (2 days/week) and then received the real intervention of TBS (iTBS 1200) over the posterior superior temporal sulcus for 4 weeks (2 days/week).
  *iTBS = intermittent theta burst stimulation
Arm/Group | Active-Active | Sham Control
Number analyzed (Participants) | 40 | 35
score on a scale
  Baseline | 20.8 (8) | 24.8 (6.9)
  During TBS | 21.9 (8.1) | 25.8 (7)
  Post TBS | 21.8 (9) | 24.8 (6.3)
  One month follow up | 22 (8.6) | 26 (7.1)

5. Secondary Outcome: Functional MRI (Biological Motion Task)
Description: The MRI data have to be pre-processed before analysis. It may take few years.
Time Frame: baseline; during TBS (4 weeks after baseline); post TBS (8 weeks after baseline)
Reporting Status: Not Posted

6. Secondary Outcome: Resting State fMRI
Description: The MRI data have to be pre-processed before analysis. It may take few years.
Time Frame: baseline; during TBS (4 weeks after baseline); post TBS (8 weeks after baseline)
Reporting Status: Not Posted

7. Secondary Outcome: Diffusion Tensor Imaging
Description: The MRI data have to be pre-processed before analysis. It may take few years.
Time Frame: baseline; during TBS (4 weeks after baseline); post TBS (8 weeks after baseline)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: The adverse event would be assessed before and after intervention every session, up to 4 weeks.
Arm/Group | Active-Active | Sham-Active
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/35
Other Adverse Events (participants affected / at risk) | 4/40 | 10/35
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active-Active (N=40) | Sham-Active (N=35)
Pain at application site (Nervous system disorders) | 4 | 0 — Phase 1
Pain at application site (Nervous system disorders) | 4 | 10 — Phase 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-14): https://cdn.clinicaltrials.gov/large-docs/89/NCT03621189/Prot_SAP_000.pdf